CLINICAL TRIAL: NCT02794415
Title: Translating Exercise Into the HIV Community: Evaluating a Community-based Exercise Intervention to Improve the Health of Adults Living With HIV
Brief Title: Evaluating a Community-Based Exercise Intervention With Adults Living With HIV: An Interrupted Time Series Study
Acronym: CBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: YMCA (Other)
Responsible Party: Principal Investigator, Kelly O'Brien, Associate Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REB Protocol #32910
Record Dates: First submitted 2016-06-01; First posted 2016-06-09 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: HIV
Keywords: HIV; disability; rehabilitation; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Community-based exercise (Other)
  Interventions: Other: Community-based exercise

INTERVENTIONS:
Other: Community-based exercise — Intervention Phase (6 months): The HIV Community-Based Exercise (CBE) intervention is a 6-month exercise program at the Central Toronto YMCA. Participants will meet the fitness instructor to establish an individualized exercise program that will include a combination of aerobic, resistive, neuromotor and flexibility training. Participants will attend exercise sessions for ~1.5 hour, 3 times per week for 24 weeks. Sessions will be supervised weekly by a fitness instructor.
  Post-Intervention Phase (8 months): At the end of the 24 week intervention, participants will be encouraged to continue to engage in unsupervised exercise 3 times per week. As per usual practice at the YMCA, a fitness instructor will be available to monitor participants monthly.

SUMMARY:
The primary aim of this research is to evaluate a community-based exercise (CBE) intervention for adults living with HIV within the community with the goal of reducing disability and enhancing health (cardiopulmonary, strength, weight and body composition, and neurocognitive outcomes) and contextual factor outcomes (social support, stigma, mastery, coping) for adults living with HIV.

DETAILED DESCRIPTION:
Investigators will use the RE-AIM Framework to evaluate the community-based exercise (CBE) intervention. The RE-AIM Framework includes criteria to evaluate the impact and translation of an intervention at both individual and organizational-levels in order to promote uptake, transferability and ultimately enhance the public health impact of health promotion interventions.

Specific study objectives are: 1) To determine the extent (proportion of sessions attended, frequency, intensity, time, type) to which adults with HIV participate in a CBE intervention; 2) To assess the effect of a CBE intervention on disability and health outcomes and intrinsic and extrinsic factor outcomes for people living with HIV; 3) To assess engagement in CBE for adults with HIV over time (adherence, level of physical activity); and 4) To evaluate the process (strengths and challenges; feasibility; accessibility, long term sustainability) of implementing a CBE intervention within the community from the perspective of recreation providers (fitness instructors; managers) and people living with HIV.

Investigators will conduct a prospective longitudinal study using mixed methods to evaluate a CBE intervention in the community with people living with HIV. They will use an interrupted time series (ITS) design in combination with qualitative interviews to assess outcomes at baseline (pre-testing phase), during (intervention phase) and after the CBE intervention (post-testing phase) to evaluate the short- and long-term effect of CBE.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older) living with HIV in Toronto who consider themselves medically stable and safe to engage in exercise and who are willing to participate in a 22 month study involving a 14 month CBE intervention at the YMCA.

Exclusion Criteria:

* Not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Maximum oxygen consumption (VO2max) | Bimonthly outcome assessment throughout baseline monitoring (8 months), intervention (6 months) and follow-up (8 months) for a total of 22 months
  Maximum oxygen consumption (VO2max) ml/kg/min

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data supporting the conclusions of this article are included within the article and its supplemental files. The data used and/or analysed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data supporting the conclusions of this article are included within the article and its supplemental files. The data used and/or analysed during the current study are available from the corresponding author on reasonable request.
Access Criteria: The data supporting the conclusions of this article are included within the article and its supplemental files. The data used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] O'Brien KK, Bayoumi AM, Solomon P, Tang A, Murzin K, Chan Carusone S, Zobeiry M, Nayar A, Davis AM. Evaluating a community-based exercise intervention with adults living with HIV: protocol for an interrupted time series study. BMJ Open. 2016 Oct 20;6(10):e013618. doi: 10.1136/bmjopen-2016-013618. PMID 27798038
- [Background] O'Brien KK, Davis AM, Chan Carusone S, Avery L, Tang A, Solomon P, Aubry R, Zobeiry M, Ilic I, Pandovski Z, Bayoumi AM. Examining the impact of a community-based exercise intervention on cardiorespiratory fitness, cardiovascular health, strength, flexibility and physical activity among adults living with HIV: A three-phased intervention study. PLoS One. 2021 Sep 24;16(9):e0257639. doi: 10.1371/journal.pone.0257639. eCollection 2021. PMID 34559851
- [Background] Solomon P, Carusone SC, Davis AM, Aubry R, O'Brien KK. Experiences of People Living With HIV in Community Based Exercise: A Qualitative Longitudinal Study. J Int Assoc Provid AIDS Care. 2021 Jan-Dec;20:2325958221995344. doi: 10.1177/2325958221995344. PMID 33611978
- [Background] Solomon P, Chan Carusone S, Davis AM, Aubry R, O'Brien KK. A Qualitative Study of Fitness Coaches' Experiences in Community Based Exercise with People Living with HIV. J Int Assoc Provid AIDS Care. 2021 Jan-Dec;20:23259582211046762. doi: 10.1177/23259582211046762. PMID 34668422
- [Derived] Turner JR, Chow J, Cheng J, Hassanali F, Sevigny H, Sperduti M, Chan Carusone S, Dagenais M, O'Brien KK. Wireless physical activity monitor use among adults living with HIV in a community-based exercise intervention study: a quantitative, longitudinal, observational study. BMJ Open. 2023 Apr 5;13(4):e068754. doi: 10.1136/bmjopen-2022-068754. PMID 37019491